CLINICAL TRIAL: NCT01465100
Title: Hepatocyte Transplantation for Phenylketonuria
Brief Title: Liver Cell Transplant for Phenylketonuria
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was funded by NIH grant; grant funding ended in June 2023 without enrollment of additional subjects; the only subject enrolled was in 2011.
Sponsor: Ira Fox (Other)
Responsible Party: Sponsor-Investigator, Ira Fox, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19030291
Record Dates: First submitted 2011-10-20; First posted 2011-11-04 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Phenylketonuria
Keywords: phenylketonuria; hepatocyte
MeSH Terms: conditions — Phenylketonurias | interventions — Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hepatocyte Transplantation (Experimental): See Below.
  Interventions: Radiation: Preparative Radiation Therapy; Procedure: Hepatocyte Transplant; Drug: Immunosuppression; Other: Liver Evaluation; Behavioral: Neuro-psychological Assessment; Diagnostic Test: Whole body Phe oxidation testing; Procedure: Liver Biopsy

INTERVENTIONS:
Radiation: Preparative Radiation Therapy — Subjects will undergo CT-based simulation and treatment planning for radiation therapy. Once a suitable hepatocyte donor is found and the cell count and viability is acceptable for transplantation, patients will receive Intensity-Modulated Radiation Therapy (IMRT) in one fraction(10 Gy)to the right lobe of the liver (but not exceeding 50% of the liver mass).
Procedure: Hepatocyte Transplant — Transplantation of hepatocytes into the liver will be through the portal vein, either accessed transhepatically, or by umbilical vein. After cell transplantation, measures will be taken to provide chronic access to the portal venous circulation system. If chronic access is achieved, patients will be seen in the PCTRC once a week to assess the site.
  Hepatocytes from more than one donor may be required to provide sufficient numbers of cells for transplantation to correct the disease process and to optimize Phe tolerance. Hepatocytes will be infused until the goal number of hepatocytes is infused. If viable hepatocytes remain after the goal number has been infused, the remaining cells will also be infused, as tolerated by the patient.
Drug: Immunosuppression — Following transplantation, patients will be treated with conventional immune suppression, as is used following whole organ liver transplantation. Patients will be followed as routinely performed following organ transplantation and also followed as would normally be performed for their PKU.
Other: Liver Evaluation — Prior to the hepatocyte transplant subjects will undergo a liver evaluation which is standard for all patients who have whole organ transplants at Children's Hospital of Pittsburgh of UPMC. The evaluation includes immunosuppression medication education, psychological assessment, bloodwork to assess blood count, blood and tissue type, blood chemistries, immune system function and certain infectious diseases, EKG, chest x-ray, and abdominal ultrasound to assess blood flow to the blood vessels in the liver. A liver biopsy may be performed if, in the clinical judgment of the investigators, the subject shows clinical signs of liver failure, or is at increased risk for liver fibrosis.
Behavioral: Neuro-psychological Assessment — Subjects will undergo a repeat neuropsychological assessment at 6, 12 and 24 months post-transplant (Visits 4 and 6 and the End of Study Visit) which will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Diagnostic Test: Whole body Phe oxidation testing — Patient will again be asked to not eat or drink for at least four hours prior to testing. Isotopic monitoring of whole body Phe oxidation will be performed pre-transplant and at every follow-up visit following the final hepatocyte infusion. An additional Phe oxidation test may also be completed in the event of suspected graft rejection.
Procedure: Liver Biopsy — Liver biopsies will be performed at 3 and 12 months post-transplant to assess for the presence of donor hepatocytes, and may be completed in the event of suspected graft rejection.

SUMMARY:
Human phenylketonuria (PKU) results from phenylalanine hydroxylase (PAH) deficiency, and represents one of the most common and extensively studied single-gene Mendelian disorders in humans. Unfortunately, optimum clinical outcome demands lifelong dietary restriction through adherence to an unpalatable and expensive artificial diet. Challenges in maintaining traditional therapy lead to increasing phenylalanine (Phe) levels in patients as they approach adulthood with an incumbent severe burden of psychosocial and intellectual difficulties. The recent introduction of the new medication Sapropterin for treatment of PKU has improved Phe control and dietary tolerance in some patients, but at enormous cost to patients and insurers for the FDA designated orphan product. Thus, there is an unmet need for novel therapies to correct PKU. PAH is almost exclusively expressed in the liver in humans. The main objective of the current proposal is to examine the safety and efficacy of hepatocyte transplantation in patients with PKU.

DETAILED DESCRIPTION:
Hepatocytes from more than one donor may be required to provide sufficient numbers of cells for transplantation to correct the disease process. We have previously estimated that the hepatic mass of a recipient approaches 4 x 10 to the 9th power hepatocytes/kg. However, this is just an estimate and the true mass may be twice this number. Our goal is to attempt to infuse at least 2x10 to the 8th power cells/kg. Once it has been determined that IND release criteria for the hepatocytes has been met, the patient will then receive Intensity-Modulated Radiation Therapy (IMRT), and the hepatocyte transplant will begin.

Preparative Liver Irradiation: A portion of the right hepatic lobe comprising between 35-50% of the entire liver volume will be irradiated to a dose of 10 Gy in a single fraction using a linear accelerator-based stereotactic radiosurgery system with intensity-modulated radiation therapy planning (IMRT). Respiratory gating will be used to further increase the accuracy of delivering the dose to a specified volume and limiting the exposure to adjacent tissues. After hepatic irradiation, the right or main portal vein will be occluded transiently (0-90 min) to provide a compensatory mitotic signal to donor hepatocytes. Transient portal vein occlusion or embolization has been shown in primates to provide the appropriate mitotic signals necessary for donor cell proliferation. At that time, donor hepatocytes will be transplanted into the irradiated portion of the recipient's liver.

The number of infusions from each donor liver will depend on the tolerance of the patient to infusion (avoidance of portal vein thrombosis and portal vein to systemic venous system shunting), and viability of donor hepatocytes. The hepatocytes from each donor liver will be given over three to four infusions, every 6 to 8 hours, until the cells are no longer viable, approximately twenty-four hours after initial preparation. Ideally, the infusion catheter will be maintained just outside the portal circulation in the umbilical vein remnant so the patient can be potentially discharged from the hospital until the next donor liver is available. Since we do not yet know from our experience the number of cells needed for transplant in order to improve function so that a metabolic disease is cured, we will continue to infuse hepatocytes as donors become available until reaching the goal volume of hepatocytes and until viability of cells has expired. Using hepatocytes from multiple donors will help to ensure that an adequate number of cells is infused while maintaining portal pressure in the normal range.Phe levels will be collected once a week by the subject, using a capillary blood sample on a newborn screening filter paper, and mailed to CHP. Phe levels will also be collected in a venous sample monthly. During months when a Follow-Up Visit is scheduled, both a venous and capillary sample will be collected.

Subjects will receive careful dietary observation post-transplant through the UPMC Children's Hospital of Pittsburgh Division of Medical Genetics research dietician. Three-day diet records will be completed once a month for six months, then every three months thereafter. Diet should remain unchanged throughout the study, unless directed by study staff.

Subjects will undergo a repeat neuropsychological assessment at 6, 12 and 24 months post-transplant (Visits 4 and 6 and the End of Study Visit) which will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.

Isotopic monitoring of whole body Phe oxidation will be performed at every follow-up visit following the final hepatocyte infusion. An additional Phe oxidation test may also be completed in the event of suspected graft rejection.

Liver biopsies will be performed at 3 and 12 months post-transplant to assess for the presence of donor hepatocytes, and may be completed in the event of suspected graft rejection.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diagnosis of classical PKU, as determined by a PAH mutation known to cause classical PKU, or a Phe >20 mg/dL at any time.
2. Patients must have poor control on standard therapy (i.e. Kuvan or diet alone) as defined by two consecutive Phe levels of > 12 mg/dL in the past six months. This is two times the recommended level. If the patient is being treated with Palynziq, they must discontinue treatment for at least two months before participating in this trial.
3. Baseline I.Q. ≥70 as assessed by Wechsler Abbreviated Scale of Intelligence (4-subtest IQ)
4. Must have a complete evaluation, including dietary records, in a PKU clinic in the past twelve months
5. Age between 14 and 55 years
6. Stated willingness to comply with all study procedures and availability for the duration of the study
7. Sexually active female subjects must agree to use two highly effective forms of contraception for the duration of the study

Exclusion Criteria:

1. I.Q. <70
2. Known biopterin synthesis defects
3. Subject has active malignancy
4. Subject has known allergy or other contraindication to immune suppression medications (and their alternatives) required post transplant for the prevention of rejection
5. Subject has sepsis, pneumonia, other active infection, or other secondary life-threatening organ dysfunction at Screening or Baseline Visits. Subject may be re-screened once infection has cleared.
6. Subject is pregnant or breastfeeding
7. Subject has positive HIV serostatus
8. Liver biopsy shows significant fibrosis, defined by the Ishak Stage 5: bridges with occasional nodules, or higher. Liver biopsy will be performed if, in the clinical judgment of the investigators, subject has clinical signs of liver failure, or increased risk of liver fibrosis.
9. Any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or not completing the required study follow-up
10. Concurrent disease or condition that would interfere with study participation or safety

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10-12 (Actual); Primary Completion 2015-08-21 (Actual); Study Completion 2016-06-17 (Actual)

PRIMARY OUTCOMES:
Improvement/reversal of characteristics of PKU | 24 months post hepatocyte transplant
  Measured as a 50% decrease in Phe from baseline study level.

SECONDARY OUTCOMES:
Engraftment of Hepatocytes | 3 months
  Liver biopsy will be performed at 3 months post-transplant to assess for the presence of donor hepatocytes, and may be completed in the event of suspected graft rejection.
Engraftment of Hepatocytes | 12 months
  Liver biopsy will be performed at 12 months post-transplant to assess for the presence of donor hepatocytes, and may be completed in the event of suspected graft rejection.
Engraftment of Hepatocytes | up to 24 months
  Laboratory tests of hepatic function
Wechsler Abbreviated Scale of Intelligence-third edition (WASI-III) | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visits 4). T-scores ranging from 20-80 with higher scores reflecting better functioning. Scores are transformed to standard scores ranging from 50-150 again with higher scores representing better functioning. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Wechsler Abbreviated Scale of Intelligence-third edition (WASI-III) | 12 months
  Subjects will undergo a repeat neuropsychological assessment at 12 months post-transplant (Visit 6) T-scores ranging from 20-80 with higher scores reflecting better functioning. Scores are transformed to standard scores ranging from 50-150 again with higher scores representing better functioning. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Wechsler Abbreviated Scale of Intelligence-third edition (WASI-III) | 24 months
  Subjects will undergo a repeat neuropsychological assessment at 24 months post-transplant (End of Study Visit) T-scores ranging from 20-80 with higher scores reflecting better functioning. Scores are transformed to standard scores ranging from 50-150 again with higher scores representing better functioning. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Delis Kaplan Executive Functioning System (D-KEFS) | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). 16 subtests. Test scores vary depending on primary interest and comparisons. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Delis Kaplan Executive Functioning System (D-KEFS) | 12 months
  Subjects will undergo a repeat neuropsychological assessment at 12 months post-transplant (Visit 6) 16 subtests. Test scores vary depending on primary interest and comparisons. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Delis Kaplan Executive Functioning System (D-KEFS) | 24 months
  Subjects will undergo a repeat neuropsychological assessment at 24 months post-transplant (End of Study Visit). 16 subtests. Test scores vary depending on primary interest and comparisons. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Connors Continuous Performance Test-third edition (CPT-III) | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). T scores ranging from <40 to 90 with higher scores reflecting worse function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Connors Continuous Performance Test-third edition (CPT-III) | 12 months
  Subjects will undergo this neuropsychological assessment at 12 months post-transplant (Visit 6). T scores ranging from <40 to 90 with higher scores reflecting worse function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Connors Continuous Performance Test-third edition (CPT-III) | 24 months
  Subjects will undergo this neuropsychological assessment at 24 months post-transplant (End of Study Visit). T scores ranging from <40 to 90 with higher scores reflecting worse function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Adaptive Behavior Assessment System-third edition (ABAS-III) | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). Subtests scaled scores range from 1-15, composite transform to standard scores ranging from 40-120. Higher scores for all reflect better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Adaptive Behavior Assessment System-third edition (ABAS-III) | 12 months
  undergo this neuropsychological assessment at 12 months post-transplant (Visit 6). Subtests scaled scores range from 1-15, composite transform to standard scores ranging from 40-120. Higher scores for all reflect better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Adaptive Behavior Assessment System-third edition (ABAS-III) | 24 months
  Subjects will undergo this neuropsychological assessment at 24 months post-transplant (End of Study Visit). Subtests scaled scores range from 1-15, composite transform to standard scores ranging from 40-120. Higher scores for all reflect better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
SF-36 Health Survey | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). scores are transformed to scale scores of 0-100 with higher scores reflecting better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
SF-36 Health Survey | 12 months
  Subjects will undergo this neuropsychological assessment at 12 months post-transplant (Visit 6). scores are transformed to scale scores of 0-100 with higher scores reflecting better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
SF-36 Health Survey | 24 months
  Subjects will undergo this neuropsychological assessment at 24 months post-transplant (End o Study Visit). scores are transformed to scale scores of 0-100 with higher scores reflecting better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Beck Depression Inventory | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). scores range from 0-63 with higher scores representing poorer function/more prominent depression. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Beck Depression Inventory | 12 months
  Subjects will undergo this neuropsychological assessment at 12 months post-transplant (Visit 6). scores range from 0-63 with higher scores representing poorer function/more prominent depression. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Beck Depression Inventory | 24 months
  Subjects will undergo this neuropsychological assessment at 24 months post-transplant (End of Study Visit). scores range from 0-63 with higher scores representing poorer function/more prominent depression. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Behavior Rating Inventory of Executive Function (BRIEF-parent version) | 6 months
  Parents of subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4) regarding the behavior of their child. scores are converted to T-scores ranging from 40-90 with higher scores representing greater dysfunction. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Behavior Rating Inventory of Executive Function (BRIEF-parent version) | 12 months
  Parents of subjects will undergo this neuropsychological assessment at 12 months post-transplant (Visit 6) regarding the behavior of their child. scores are converted to T-scores ranging from 40-90 with higher scores representing greater dysfunction. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Behavior Rating Inventory of Executive Function (BRIEF-parent version) | 24 months
  Parents of subjects will undergo this neuropsychological assessment at 24 months post-transplant (End of Study Visit) regarding the behavior of their child. scores are converted to T-scores ranging from 40-90 with higher scores representing greater dysfunction. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Behavior Assessment System for Children-second edition (BASC-II) | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). Scores converted to T-scores 40-90 with higher scores representing poorer function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Behavior Assessment System for Children-second edition (BASC-II) | 12 months
  Subjects will undergo this neuropsychological assessment at 12 months post-transplant (Visit 6). Scores converted to T-scores 40-90 with higher scores representing poorer function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Behavior Assessment System for Children-second edition (BASC-II) | 24 months
  Subjects will undergo this neuropsychological assessment at 24 months post-transplant (End of Study Visit). Scores converted to T-scores 40-90 with higher scores representing poorer function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Child Health Questionnaire (CHQ) | 6 months
  Subjects will undergo this neuropsychological assessment at 6 months post-transplant (Visit 4). Scores converted to a 0-100 scale with higher scores evidencing better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Child Health Questionnaire (CHQ) | 12 months
  Subjects will undergo this neuropsychological assessment at 12 months post-transplant (Visit 6). Scores converted to a 0-100 scale with higher scores evidencing better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.
Child Health Questionnaire (CHQ) | 24 months
  Subjects will undergo this neuropsychological assessment at 24 months post-transplant (End of Study Visit). Scores converted to a 0-100 scale with higher scores evidencing better function. Results will be compared to results obtained pre-transplant to determine whether an improvement in assessment scoring is associated with the transplant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ira J Fox, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No